CLINICAL TRIAL: NCT02523300
Title: Prognostic Value of Single-dose Glucocorticoid After Endovascular Repair for Aortic Dissection
Brief Title: Glucocorticoid on the Prognosis of TEVAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zaiping JING, Director of Vascular Surgery Department, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GC-AD-2015-07
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection | interventions — Endovascular Aneurysm Repair; Glucocorticoids; Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEVAR+GC (Experimental): The patients underwent TEVAR. Then glucocorticoids will be intravenously given after TEVAR
  Interventions: Procedure: TEVAR; Drug: Glucocorticoids
- TEVAR+Vehicle (Placebo Comparator): The patients underwent TEVAR. Then saline will be given after TEVAR
  Interventions: Procedure: TEVAR; Drug: saline

INTERVENTIONS:
Procedure: TEVAR — The patients will be undertaken TEVAR
  Other Names: thoracic endovascular aortic repair
Drug: Glucocorticoids — About 120 patients will be given glucocorticoids within 2h after TEVAR as experimental group
  Other Names: methylprednisolone
  Arms: TEVAR+GC
Drug: saline — The other 120 patients will be given saline as control group
  Other Names: Vehicle
  Arms: TEVAR+Vehicle

SUMMARY:
To explore the potential prognostic effect of glucocorticoid on the postoperative aorta-related adverse events after aortic dissections patients underwent thoracic endovascular aortic repair (TEVAR), glucocorticoid (30mg/kg) will be intravenously given within 2h after TEVAR.

DETAILED DESCRIPTION:
This is a prospective, open, single-center, randomized controlled trial. Number of patients: 240 patients will be included and undertaken TEVAR.About 120 patients will be given glucocorticoid within 2h after TEVAR as experimental group, and the other 120 patients will be given saline as control group.

Follow-up: 1. aortic computed tomographic angiography (CTA) examination 6, 12 and 24 months after TEVAR; 2. telephone or clinical follow-up at 1, 2, 3, 6, 12 and 24 months.

Primary outcome measure: aorta-related adverse events. Second outcome measure: 30-day mortality after TEVAR, success rate of endovascular repair, drug-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. age from 18 to 80, male or unpregnant female;
2. diagnosed as aortic dissection, excluding intramural hematoma and penetrating aortic ulcer;
3. complicated aortic dissection with definite indications of TEVAR;
4. voluntarily signed the informed consent form;
5. good compliance with the instructions and cooperate with follow-up.

Exclusion Criteria:

1. no appropriate vessel approaches;
2. patients with connective tissue diseases (such as Marfan syndrome);
3. patients with endocrine disease,such as diabetes mellitus, or undergoing hormonotherapy;
4. bad compliance with the instructions and follow-up;
5. allergic to nitinol and contrast medium;
6. estimated life expectancy is less than 24 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Aorta-related adverse events | 24 months

SECONDARY OUTCOMES:
30-day mortality after TEVAR | 30 days
Success rate of endovascular repair | 24 months
Drug-related adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Zaiping Jing, Doctor, Principal Investigator — Department of Vascular Surgery, Changhai Hospital

REFERENCES:
- [Derived] Wu M, Zhang L, Bao J, Zhao Z, Lu Q, Feng R, Song C, Zhou J, Jing Z. Postoperative glucocorticoid enhances recovery after endovascular aortic repair for chronic type B aortic dissection: a single-center experience. BMC Cardiovasc Disord. 2016 Mar 25;16:59. doi: 10.1186/s12872-016-0234-2. PMID 27013022